CLINICAL TRIAL: NCT05871489
Title: Strengthening Evidence on Optimal Multidrug-resistant Tuberculosis Treatment Regimens Through Improved Epidemiologic Methods
Brief Title: Strengthening Evidence on Optimal Multidrug-resistant Tuberculosis Treatment Regimens
Acronym: STEM-TB
Status: Active, not recruiting | Type: Observational
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Partners in Health (Other); Socios En Salud Sucursal, Peru (Other)
Responsible Party: Principal Investigator, Molly Franke, Associate Professor of Global Health and Social Medicine, Harvard Medical School (HMS and HSDM)
Other Study IDs: R01AI146095 (NIH); R01AI146095 (NIH)
Record Dates: First submitted 2023-05-01; First posted 2023-05-23 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-06

CONDITIONS: Tuberculosis, Multidrug-Resistant; HIV
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Lesotho Cohort: 200 patients receiving an all-oral shorter regimen in Lesotho under routine program conditions.
  Interventions: Drug: Bdq, Lzd, Lfx, Dlm, Cfz (9-12 months)
- Peru Cohort: 50 patients receiving an all-oral shorter regimen in Peru under routine program conditions.
  Interventions: Drug: Bdq, Lzd, Lfx, Dlm, Cfz (9-12 months)
- Kazakhstan Cohort: 550 patients receiving an all-oral shorter regimen in Kazakhstan under routine program conditions.
  Interventions: Drug: Bdq, Lzd, Lfx, Dlm, Cfz (9-12 months); Drug: Bdq, Lzd, Lfx, Cfz, Cs (9-12 months); Drug: Bdq, Lzd, Lfx, Z, Dlm (9-12 months)

INTERVENTIONS:
Drug: Bdq, Lzd, Lfx, Dlm, Cfz (9-12 months) — Bdq, Lzd, Lfx, Dlm, Cfz for nine months, with extension to 12 months as needed
Drug: Bdq, Lzd, Lfx, Cfz, Cs (9-12 months) — Bdq, Lzd, Lfx, Cfz, Cs for nine months, with extension to 12 months as needed
  Groups: Kazakhstan Cohort
Drug: Bdq, Lzd, Lfx, Z, Dlm (9-12 months) — Bdq, Lzd, Lfx, Z, Dlm for nine months, with extension to 12 months as needed
  Groups: Kazakhstan Cohort

SUMMARY:
This is a multisite prospective cohort study of patients with multidrug- or rifampin-resistant tuberculosis who are treated with an all-oral shortened regimen under routine program conditions in one of three countries (Peru, Lesotho, Kazakhstan).

ELIGIBILITY:
Inclusion Criteria:

* All patients with pulmonary tuberculosis that is resistant to rifampin (RIF) or to both RIF and isoniazid who initiate an all-oral treatment regimen (short or long) under routine or operational conditions, per local country guidance, will be included.

Exclusion Criteria:

* Exclusions are based on local guidance in each country. Currently, individuals with fluoroquinolone resistant tuberculosis are excluded from all-oral shortened treatment.

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will prospectively follow an observational cohort patients with confirmed MDR-TB who initiate one of the following MDR-TB regimens of interest: (1) an individualized 18-24 month all-oral regimen containing BDQ and/or DLM, designed according to 2019 WHO guidance (Lesotho); or (2) a standardized, shortened all-oral regimen containing BDQ or DLM.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
End-of-treatment outcome | 9-12 months after treatment initiation
  Number of individuals experiencing each tuberculosis treatment outcome (cure, completion, death, failure, lost-to-follow-up), assessed at the end of treatment by a clinician, based on culture results
Final tuberculosis treatment outcome | 6-24 months after treatment completion
  Number of individuals experiencing each final tuberculosis treatment outcome (cure, completion, death, failure, lost-to-follow-up, relapse), assessed at 6, 12, and 24 months by a clinician, based on culture results
Adverse events of interest | Tuberculosis treatment, an average of 9 months
  Assessed by a clinician based on symptomatology, subjective screening, and/or laboratory findings

CONTACTS AND LOCATIONS:
Locations (3):
- Partners In Health, Kazakhstan, Almaty, Kazakhstan
- Partners In Health, Lesotho, Maseru, Lesotho
- Socios En Salud, Lima, Lima Province, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rashitov M, Franke MF, Trevisi L, Bekbolatova G, Shalimova J, Eshmetov G, Bektasov S, LaHood A, Arlyapova N, Osso E, Yedilbayev A, Korotych O, Ciobanu A, Skrahina A, Mitnick CD, Seung KJ, Algozhin Y, Rich ML. Safety and Effectiveness of 3 Novel All-Oral Shortened Regimens for Rifampicin- or Multidrug-Resistant Tuberculosis in Kazakhstan. Clin Infect Dis. 2024 Oct 15;79(4):1046-1053. doi: 10.1093/cid/ciae305. PMID 38833593